CLINICAL TRIAL: NCT05808114
Title: Quality of Life in Children With Psychiatric Disorders and Parental Well-being: Effects of Group CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Sarianna Barron-Linnankoski, Principal Investigator, Helsinki University Central Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUS/2699/2018
Record Dates: First submitted 2023-03-15; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Quality of Life
Keywords: Quality of life; Health-related quality of life; Children; cognitive behavioral therapy; group cognitive behavioral therapy; parental wellbeing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group cognitive behavioral therapy (Experimental): Friends Program
  Interventions: Behavioral: Friends program
- Treatment as Usual (Experimental): A TAU condition during which participants received routine care services tailored to each child individually.
  Interventions: Behavioral: TAU

INTERVENTIONS:
Behavioral: Friends program — A GCBT intervention comprising ten weekly 60-minute sessions followed by two booster sessions
  Arms: Group cognitive behavioral therapy
Behavioral: TAU — Individually tailored and delivered specialized child psychiatric care
  Arms: Treatment as Usual

SUMMARY:
This study examines the immediate and long-term effectiveness of a group cognitive behavioral therapy intervention (GCBT) in improving health-related quality of life (HRQOL) in children treated for mixed psychiatric disorders in naturalistic child psychiatric outpatient settings. The effects of a treatment-as-usual condition (TAU) is also examined. Further, the study aims to explore the associations among children´s HRQOL dimensions and parental well-being, and how GCBT may influence these associations.

DETAILED DESCRIPTION:
The effectiveness of GCBT and TAU at the different time points are measured using nonparametric tests, such as Friedman tests and Wilcoxon tests. The associations among children´s HRQOL dimensions and parental well-being variables at different time points are explored using a network analysis approach.

ELIGIBILITY:
Inclusion Criteria:

* child psychiatric outpatient care
* sufficient skills to participate in group sessions

Exclusion Criteria:

* child psychiatric inpatient care
* acute suicidality
* excessive physical aggression

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 109 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in self-and parent-rated health-related quality of life after the group cognitive behavior therapy (GCBT) intervention | Before and after the group cognitive behavioral intervention (duration from pre-GCBT to post-GCBT circa 4.7 months), and at a 7-month follow-up
  Children´s health-related quality of life measured using the KINDL-R measure, total scores range from 0-100 with higher scores indicating better health-related quality of life
Changes in self-and parent-rated health-related quality of life after treatment as usual (TAU) | Before and after TAU (duration circa 3.2 months)
  Children´s health-related quality of life measured using the KINDL-R measure, total scores range from 0-100 with higher scores indicating better health-related quality of life

SECONDARY OUTCOMES:
Associations among children´s health-related quality of life and parental well-being dimensions | Before and after the group cognitive behavioral intervention (duration from pre-GCBT to post-GCBT circa 4.7 months), and at a 7-month follow-up
  Children´s health-related quality of life measured using the KINDL-R measure, total scores range from 0-100 with higher scores indicating better health-related quality of life
Associations among children´s HRQOL and parental well-being dimensions (parental psychological distress) | Before and after the group cognitive behavioral intervention (duration from pre-GCBT to post-GCBT circa 4.7 months), and at a 7-month follow-up
  Parental psychological distress measured using five items of the 12-item General Health Questionnaire. The sum of the items range from 5-20 with higher scores indicating greater psychological distress
Associations among children´s HRQOL and parental well-being dimensions (parental sleep disturbance) | Before and after the group cognitive behavioral intervention (duration from pre-GCBT to post-GCBT circa 4.7 months), and at a 7-month follow-up
  Parental sleep disturbance measured using the four- item Jenkins Sleep Questionnaire. Scores range from 0-20 with higher scores indicating greater sleep disturbance